CLINICAL TRIAL: NCT00102687
Title: A Multicenter, Randomized, Open-Label Study Comparing Three Alternative Dosing Regimens of Subcutaneous Azacitidine Plus Best Supportive Care for the Treatment of Myelodysplastic Syndromes
Brief Title: Alternative Dosing Regimens of Subcutaneous Azacitidine for Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZA PH US 2004 CL003
Record Dates: First submitted 2005-01-31; First posted 2005-02-01 (Estimated); Results first posted 2010-05-28 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Aza-5 (Experimental): Azacitidine administered subcutaneously at 75mg/m^2 for 5 days on a 28 day cycle.
  Interventions: Drug: azacitidine
- Aza-5-2-2 (Experimental): Azacitidine administered subcutaneously at 75mg/m^2 for 5days with 2 days off, then for an additional 2 days, on a 28 day cycle.
  Interventions: Drug: azacitidine
- Aza-5-2-5 (Experimental): Azacitidine administered subcutaneously at 50mg/m^2 for 5 days with 2 days off, then for an additional 5 days, on a 28 day cycle.
  Interventions: Drug: azacitidine
- Maintenance Aza 5 days q 4 weeks (Experimental): Azacitidine administered subcutaneously at 75mg/m^2 for 5 days every 4 weeks.
  Interventions: Drug: azacitidine
- Maintenance Aza 5 days q 6 weeks (Experimental): Azacitidine administered subcutaneously at 75mg/m^2 for 5 days every 6 weeks.
  Interventions: Drug: azacitidine

INTERVENTIONS:
Drug: azacitidine — Azacitidine is administered subcutaneously
  Total of 18 cycles on treatment or early discontinuation.

SUMMARY:
The purpose of this study is to determine if azacitidine, combined with Best Supportive Care (BSC), is effective in treating myelodysplastic syndromes (MDS) when given according to a different doses and dosing schedules.

DETAILED DESCRIPTION:
Comparison/Control Interventions: The comparison is azacitidine at different doses and schedules.

Duration of Intervention: Treatment lasted for a maximum of 18 cycles, which is up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractory anemia, refractory anemia with ringed sideroblasts and at least one of the following: a)Anemia with hemoglobin <110g/L and requires at least 1 unit packed red blood cell transfusions every 28 days; b)Thrombocytopenia with platelet counts <100 x 10^9/L; or c)Neutropenia with absolute neutrophil count <1.5 x 10^9/L.
* OR, Refractory anemia with excess blasts or refractory anemia with excess blast in transformation, according to the French-American-British classification system for MDS.
* At least 18 years of age.
* Have a life expectancy of >7 months.
* Unlikely to proceed to bone marrow or stem cell transplantation therapy following remission.
* Have serum bilirubin levels less than or equal to 1.5 times the upper limit of the normal (ULN) range for the laboratory.
* Have serum glutamic-oxaloacetic transaminase (aspartate aminotransferase) or serum glutamic-pyruvic transaminase (alanine aminotransferase) levels less than or equal to 2 x ULN.
* Have serum creatinine levels less than or equal to 1.5 x ULN.

Exclusion Criteria:

* Secondary MDS.
* Prior treatment with azacitidine.
* Any prior history of Acute Myeloid Leukemia (AML).
* Malignant or metastatic disease within the previous 12 months.
* Uncorrected red cell folate deficiency or vitamin B12 deficiency.
* Hepatic tumors.
* Radiation, chemotherapy, or cytotoxic therapy for non-MDS conditions in the previous 12 months.
* Known or suspected hypersensitivity to azacitidine or mannitol.
* Prior transplantation or cytotoxic therapy to treat MDS. Prior use of Revlimid and Thalomid allowed after 30 day washout.
* Serious medical illness likely to limit survival to less than or equal to 7 months.
* Treatment with androgenic hormones during the previous 14 days
* Active viral infection with known human immunodeficiency virus or vial hepatitis Type B or C.
* Treatment with other investigational drugs with the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2008-08-01 (Actual); Study Completion 2008-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CL Beach, Study Director — Celgene Corporation
Locations (31):
- United States (31):
  - Comprehensive Blood and Cancer Center, Research Department, Bakersfield, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Cancer Center of Colorado Springs, The Oncology Clinic, PC, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Florida Cancer Institute, New Port Richey, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Oncology/Hematology Associates of Central Illinois, PC, Peoria, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Hematology & Oncology Specialists LLC, Metairie, Louisiana
  - Great Lakes Cancer Institute Breslin Cancer Center, Lansing, Michigan
  - The Center for Cancer Care and Research, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Oncology Services of Aberdeen, Aberdeen, South Dakota
  - Avera Cancer Institute Leukemia-Bone Marrow Transplant Center, Sioux Falls, South Dakota
  - McLeod Cancer and Blood Center, Johnson City, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology, P.A., Bedford, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, PA, Fort Worth, Texas
  - San Antonio Tumor & Blood Clinic, Fredericksburg, Texas
  - Cancer Care Centers of South Texas - HOAST, San Antonio, Texas
  - Virginia Oncology Associates - Lake Wright Cancer Center, Norfolk, Virginia
  - Highline Medical Oncology, Burien, Washington
  - Puget Sound Cancer Center, Edmonds, Washington
  - Puget Sound Cancer Center, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington

REFERENCES:
- [Background] R. Lyons, et al. Rapid onset of effectiveness with three alternative azacitidine (aza) dosing regimens in patients (pts) with myelodysplastic syndromes (MDS). Haematologica 2008;93(suppl 1):Abs.0232.
- [Background] Lyons R, et al. Tolerability and hematologic improvement assessed using three alternative dosing schedules of azacitidine in patients with myelodysplastic syndromes. Presented at the 2007 ASCO Annual Meeting, June 1-5, 2007, Chicago, IL. Abstract No. 7083
- [Background] Komrokji R, Swern AS, Grinblatt D, Lyons RM, Tobiasson M, Silverman LR, Sayar H, Vij R, Fliss A, Tu N, Sugrue MM. Azacitidine in Lower-Risk Myelodysplastic Syndromes: A Meta-Analysis of Data from Prospective Studies. Oncologist. 2018 Feb;23(2):159-170. doi: 10.1634/theoncologist.2017-0215. Epub 2017 Nov 8. PMID 29118268

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred and eighty-four patients were screened.
Groups:
- Aza-5-2-2: Azacitidine administered subcutaneously at 75mg/m^2 for 5 days with 2 days off, then for an additional 2 days, on a 28 day cycle.
- Maintenance Aza 5 Days q 4 Weeks: Azacitidine administered subcutaneously at 75mg/m^2 for 5 days every 4 weeks from month 7 to month 23
- Maintenance Aza 5 Days q 6 Weeks: Azacitidine administered subcutaneously at 75mg/m^2 for 5 days every 6 weeks from month 7 to month 23
Period: Initial Period
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5 | Maintenance Aza 5 Days q 4 Weeks | Maintenance Aza 5 Days q 6 Weeks
Started | 50 | 50 | 51 (3 randomized participants did not receive treatment.) | 0 | 0
Completed | 32 | 22 | 25 | 0 | 0
Not Completed | 18 | 28 | 26 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 3 | 5 | 0 | 0
Not completed — Adverse Event | 4 | 7 | 9 | 0 | 0
Not completed — Transformation to AML (blast > 30%) | 1 | 3 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 2 | 9 | 6 | 0 | 0
Not completed — Sponsor's decision | 0 | 1 | 1 | 0 | 0
Not completed — Failed Treatments (relapse,disease prog) | 4 | 4 | 2 | 0 | 0
Not completed — Death | 1 | 1 | 1 | 0 | 0
Period: Maintenance Period
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5 | Maintenance Aza 5 Days q 4 Weeks | Maintenance Aza 5 Days q 6 Weeks
Started | 13 (Remained on initial treatment in the maintenance period.) | 6 (Remained on initial treatment in the maintenance period.) | 8 (Remained on initial treatment in the maintenance period.) | 22 (Second randomization to one of two maintenance regimens) | 21 (Second randomization to one of two maintenance regimens)
Completed | 6 | 2 | 2 | 12 | 8
Not Completed | 7 | 4 | 6 | 10 | 13
Not completed — Withdrawal by Subject | 4 | 0 | 2 | 3 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 3
Not completed — Transformation to AML (blast > 30%) | 0 | 1 | 0 | 2 | 0
Not completed — Failed Treatment (relapse,disease prog) | 1 | 1 | 1 | 3 | 4
Not completed — Death | 0 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 1 | 2 | 3 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5 | Total
Number analyzed (Participants) | 50 | 50 | 51 | 151
Age, Continuous [Median (Full Range); unit: years] | 76.0 [47 to 93] | 73.0 [37 to 88] | 76.0 [54 to 91] | 75.0 [37 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 14 | 53
  Male | 33 | 28 | 37 | 98
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 47 | 41 | 48 | 136
  Black or African American | 0 | 4 | 2 | 6
  Asian/Oriental | 1 | 0 | 0 | 1
  Hispanic | 2 | 5 | 1 | 8
  Other | 0 | 0 | 0 | 0
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  Participants
    0=Fully active | 12 | 19 | 14 | 45
    1=Restricted | 32 | 23 | 29 | 84
    2=Ambulatory/capable of self care | 3 | 5 | 7 | 15
    3=Capable/limited care | 3 | 3 | 1 | 7
FAB Classification [Count of Participants; unit: Participants] — The French-American-British (FAB) classification systems refers to a series of classifications of hematologic diseases. RA = Refractory anemia; RARS = Refractory anemia with ringed sideroblasts; RAEB = Refractory anemia with excess blasts; RAEB-T = Refractory anemia with excess blasts in transformation; CMMoL = Chronic myelomonocytic leukemia; AML = Acute myelogenous leukemia
  Participants
    RA | 22 | 22 | 21 | 65
    RARS | 7 | 7 | 7 | 21
    RAEB | 14 | 14 | 17 | 45
    RAEB-T | 2 | 1 | 1 | 4
    CMMoL with <5% blasts | 3 | 3 | 1 | 7
    CMMoL with >=5% blasts | 2 | 1 | 1 | 4
    CMMoL with missing blasts | 0 | 2 | 3 | 5
    AML | 0 | 0 | 0 | 0
    Other | 0 | 0 | 0 | 0
Transfusion Dependence - Platelets [Count of Participants; unit: Participants] — Does the participant's disease cause them to be dependent upon transfusions of platelets?
  Participants
    Platelet transfusion dependent | 4 | 2 | 1 | 7
    Not platelet transfusion dependent | 46 | 48 | 50 | 144
Transfusion Dependence Status - RBCs [Count of Participants; unit: Participants] — Does the participant's disease cause them to be dependent upon transfusions of red blood cells (RBCs)?
  Participants
    RBC transfusion dependent | 25 | 24 | 22 | 71
    Not RBC transfusion dependent | 25 | 26 | 29 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants In Best Hematological Response Categories as Determined by the Investigator Using International Working Group 2000 (IWG 2000) Criteria For Myelodysplastic Syndromes (MDS) During the Initial Study Period.
Description: Participant counts by best hematological response; complete remission(CR) is better than a partial remission(PR) which is better than stable disease(SD).
  Investigator determined responses followed IWG 2000 criteria for MDS CR: repeat bone marrow show <5% myeloblasts, and peripheral blood evaluations lasting >=2 months of hemoglobin(>110 g/L), neutrophils(>=1.5x10^9/L), platelets(>=100x10^9/L), blasts (0%) and no dysplasia PR is the same as CR for peripheral blood: bone marrow shows blasts decrease by >=50% or a less advanced FAB classification from pretreatment (see Population Descrip)
Time Frame: Day 1 (randomization) to 6 months
Population: Intent to treat population. Patients without a second bone marrow assessment could not be evaluated for hematologic response.
  (Outcome Description continued)SD is a failure to achieve at least a PR, but with no evidence of progression for at least 2 months.
Measure: Number; unit: participants
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5
Number analyzed (Participants) | 50 | 50 | 51
participants
  Overall Response (CR+PR) | 4 | 3 | 4
  Complete remission (CR) | 2 | 2 | 2
  Partial remission (PR) | 2 | 1 | 2
  Stable disease | 22 | 19 | 20

2. Primary Outcome: Number of Participants With Best Hematological Improvement Derived Using International Working Group 2000 (IWG 2000) Criteria for MDS During the Initial Study Period.
Description: IWG 2000 Criteria: Pretreatment=hemoglobin <110g/L or RBC transfusion-dependence, platelet count <100x10^9/L or platelet transfusion dependence, absolute neutrophil count <1.5x10^9/L.
  Erythroid response: Major->20g/L increase in hemoglobin or transfusion independence. Minor- 10-20g/L increase in hemoglobin or >=50% decrease in transfusion requirements.
  Platelet response: Major-absolute increase of platelet count by >=30x10^9/L or platelet transfusion independence. Minor->=50% increase in platelet count with net increase >10x10^9/L but <30x10^9/L.
  (continued in Population Description)
Time Frame: Day 1 (randomization) to 6 months
Population: Intent to treat population. Patients count only once for best response within an improvement category.
  (Outcome Description continued) Neutrophil response: Major->=100% increase in neutrophil count or an absolute increase of >0.5x10^9/L. Minor->=100% increase but an absolute increase of <0.5x10^9/L.
Measure: Number; unit: participants
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5
Number analyzed (Participants) | 50 | 50 | 51
participants
  Any Improvement n=50,49,47 | 29 | 20 | 26
  Erythroid response - Major n=44,43,41 | 18 | 15 | 18
  Erythroid response - Minor n=44,43,41 | 4 | 1 | 2
  Platelet response - Major n=24,28,28 | 10 | 11 | 10
  Platelet response - Minor n=24,28,28 | 2 | 0 | 0
  Neutrophil response - Major n=24,22,16 | 4 | 3 | 3
  Neutrophil response - Minor n=24,22,16 | 2 | 0 | 0

3. Primary Outcome: Number of Participants With Overall Best Hematologic Response and Hematologic Improvement Based on IWG 2000 Criteria For MDS During the Initial Study Period
Description: Number of participants whose best hematological outcome was either complete remission (CR), partial remission (PR) (as determined by the investigator), or any hematologic improvement (based on the IWG 2000 criteria for MDS). See previous outcomes for detailed definitions.
Time Frame: Day 1 (randomization) to 6 months
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5
Number analyzed (Participants) | 50 | 50 | 51
participants | 30 | 20 | 27

4. Secondary Outcome: Baseline Hemoglobin Values
Description: The median values for hemoglobin based on blood tests performed on study day 1 (prior to study treatment) constitute a baseline measure for hemoglobin. Baseline values are used to compare to values following treatment.
Time Frame: Day 1 (randomization)
Population: Intent to treat population
Measure: Median (Full Range); unit: g/L
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5
Number analyzed (Participants) | 50 | 49 | 50
g/L | 94.0 [63.0 to 131.0] | 98.0 [70.0 to 135.0] | 95.5 [59.0 to 145.0]

5. Secondary Outcome: Change From Baseline in Hemoglobin at End of Initial Study Period (6 Months)
Description: The difference between hemoglobin values at the end of the initial study period minus the hemoglobin values at baseline.
Time Frame: 6 months
Population: Intent to treat population
Measure: Median (Full Range); unit: g/L
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5
Number analyzed (Participants) | 50 | 49 | 46
g/L | 2.3 [-25.9 to 41.8] | 2.9 [-33.0 to 31.7] | 5.3 [-20.4 to 30.4]

6. Primary Outcome: Number of Participants Who Improved or Maintained The Hematologic Response From the Initial Study Period (Based on IWG 2000 Criteria For MDS) During the Maintenance Period
Description: Hematologic response during the maintenance period are compared to the response in the initial study period. Initial response could have been a complete remission, a partial remission, stable disease or a hematologic improvement. Maintenance period best response is after randomization to a maintenance arm for those randomized, and is after the start of cycle 7 for those remaining on initial period treatment throughout the study.
Time Frame: 24 months
Population: Intent to treat population.
Measure: Number; unit: participants
Groups:
- Initial Period Treatment Continued Into Maintenance: Combines participants who continued their original treatment assigned during the initial study period through month 7 to month 23.
Arm/Group | Maintenance Aza 5 Days q 4 Weeks | Maintenance Aza 5 Days q 6 Weeks | Initial Period Treatment Continued Into Maintenance
Number analyzed (Participants) | 22 | 21 | 27
participants
  Improved response from initial study period | 7 | 10 | 12
  Maintained response from initial study period | 6 | 5 | 10

7. Secondary Outcome: Change From Baseline in Hemoglobin at the End of the Maintenance Study Period
Description: The difference between hemoglobin values at the end of the maintenance study period minus the hemoglobin values at baseline.
Time Frame: 24 months
Population: Intent to treat population
Measure: Median (Full Range); unit: g/L
Arm/Group | Maintenance Aza 5 Days q 4 Weeks | Maintenance Aza 5 Days q 6 Weeks | Initial Period Treatment Continued Into Maintenance
Number analyzed (Participants) | 22 | 21 | 26
g/L | 5.9 [-27.9 to 54.8] | 7.3 [-14.4 to 55.5] | 14.5 [-5.5 to 60.4]

8. Secondary Outcome: Baseline Platelet Values
Description: The median values for platelets based on blood tests performed on study day 1 (prior to study treatment) constitute a baseline measure for platelets. Baseline values are used to compare to values following treatment.
Time Frame: Day 1 (randomization)
Population: Intent to treat population
Measure: Median (Full Range); unit: x10(9)/L
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5
Number analyzed (Participants) | 49 | 49 | 49
x10(9)/L | 110.0 [9.0 to 516.0] | 90.0 [8.0 to 581.0] | 86.0 [8.0 to 699.0]

9. Secondary Outcome: Change From Baseline in Platelets at the End of Initial Study Period (6 Months)
Description: The difference between platelet values at the end of the initial study period minus the platelet values at baseline.
Time Frame: 6 months
Population: Intent to treat population
Measure: Median (Full Range); unit: x10^9/L
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5
Number analyzed (Participants) | 49 | 49 | 45
x10^9/L | 4.8 [-116.3 to 179.1] | 5.7 [-145.6 to 192.6] | 12.6 [-300.9 to 213.6]

10. Secondary Outcome: Change From Baseline in Platelets at the End of the Maintenance Study Period (Month 24)
Description: The difference between platelet values at the end of the maintenance study period minus the platelet values at baseline.
Time Frame: 24 months
Population: Intent to treat population
Measure: Median (Full Range); unit: x10^9/L
Arm/Group | Maintenance Aza 5 Days q 4 Weeks | Maintenance Aza 5 Days q 6 Weeks | Initial Period Treatment Continued Into Maintenance
Number analyzed (Participants) | 22 | 21 | 26
x10^9/L | 19.8 [-157.5 to 129.6] | 7.7 [-279.8 to 166.3] | 17.3 [-124.7 to 223.3]

11. Secondary Outcome: Baseline Absolute Neutrophil Count (ANC) Values
Description: The median values for ANC based on blood tests performed on study day 1 (prior to study treatment) constitute a baseline measure for ANC. Baseline values are used to compare to values following treatment.
Time Frame: Day 1 (randomization)
Population: Intent to treat population
Measure: Median (Full Range); unit: x10^9/L
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5
Number analyzed (Participants) | 50 | 49 | 50
x10^9/L | 1.6 [0.1 to 13.9] | 1.9 [0.1 to 162.3] | 2.3 [0.3 to 139.3]

12. Secondary Outcome: Change From Baseline in Absolute Neutrophil Count (ANC) at the End of Initial Study Period (6 Months)
Description: The difference between ANC values at the end of the initial study period minus the ANC values at baseline.
Time Frame: 6 months
Population: Intent to treat population
Measure: Median (Full Range); unit: x10^9/L
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5
Number analyzed (Participants) | 50 | 49 | 46
x10^9/L | -0.3 [-4.6 to 1.9] | -0.3 [-35.9 to 1.4] | -0.4 [-9.7 to 8.5]

13. Secondary Outcome: Change From Baseline in Absolute Neutrophil Count (ANC) at the End of the Maintenance Study Period (Month 24)
Description: The difference between ANC values at the end of the maintenance study period minus the ANC values at baseline.
Time Frame: 24 months
Population: Intent to treat population
Measure: Median (Full Range); unit: x10^9/L
Groups:
- Initial Period Treatment Continued Into Maintenance: Combines participants who continued their treatment assigned during the initial study period through month 7 to month 23.
Arm/Group | Maintenance Aza 5 Days q 4 Weeks | Maintenance Aza 5 Days q 6 Weeks | Initial Period Treatment Continued Into Maintenance
Number analyzed (Participants) | 22 | 21 | 26
x10^9/L | -0.1 [-17.6 to 2.0] | -0.2 [-3.1 to 1.9] | -0.4 [-19.0 to 2.3]

14. Secondary Outcome: Red Blood Cell (RBC) Transfusion Status at Baseline and End of Initial Study Period (6 Months)
Description: Shift table comparing the RBC transfusion status of patients at the end of the initial study period to the transfusion status at baseline.
Time Frame: 6 months
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5
Number analyzed (Participants) | 50 | 50 | 51
participants
  Baseline Dependent(n=25,24,22) - 6 mo Independent | 16 | 14 | 13
  Baseline Dependent(n=25,24,22) - 6 mo Dependent | 9 | 10 | 9
  Baseline Independent(n=25,26,29)- 6 mo Independent | 19 | 16 | 19
  Baseline Independent(n=25,26,29) - 6 mo Dependent | 6 | 10 | 10

15. Secondary Outcome: Platelet Transfusion Status at Baseline and End of Initial Study Period (6 Months)
Description: Shift table comparing the platelet transfusion status of patients at the end of the initial study period to the transfusion status at baseline.
Time Frame: 6 months
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5
Number analyzed (Participants) | 50 | 50 | 51
participants
  Baseline Dependent (n=4,2,1) - 6 mo Independent | 3 | 2 | 0
  Baseline Dependent (n=4,2,1) - 6 mo Dependent | 1 | 0 | 1
  Baseline Independent(n=46,48,50)- 6 mo Independent | 43 | 42 | 41
  Baseline Independent (n=46,48,50) - 6 mo Dependent | 3 | 6 | 9

16. Secondary Outcome: Red Blood Cell (RBC) Transfusion Status at Baseline and End of Maintenance Study Period (24 Months)
Description: Shift table comparing the RBC transfusion status of patients at the end of the maintenance study period to the transfusion status at baseline.
Time Frame: 24 months
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Maintenance Aza 5 Days q 4 Weeks | Maintenance Aza 5 Days q 6 Weeks | Initial Period Treatment Continued Into Maintenance
Number analyzed (Participants) | 22 | 21 | 27
participants
  Baseline Dependent (n=6,12,12) - 24 mo Independent | 5 | 12 | 10
  Baseline Dependent (n=6,12,12) - 24 mo Dependent | 1 | 0 | 2
  Baseline Independent(n=16,9,15)- 24 mo Independent | 15 | 9 | 15
  Baseline Independent (n=16,9,15) - 24 mo Dependent | 1 | 0 | 0

17. Secondary Outcome: Platelet Transfusion Status at Baseline and End of Maintenance Study Period (24 Months)
Description: Shift table comparing the platelet transfusion status of patients at the end of the maintenance study period to the transfusion status at baseline.
Time Frame: 24 months
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Maintenance Aza 5 Days q 4 Weeks | Maintenance Aza 5 Days q 6 Weeks | Initial Period Treatment Continued Into Maintenance
Number analyzed (Participants) | 22 | 21 | 27
participants
  Baseline Dependent (n=1,1,2) - 24 mo Independent | 1 | 1 | 2
  Baseline Dependent (n=1,1,2) - 24 mo Dependent | 0 | 0 | 0
  Baseline Independent(n=21,20,25)-24 mo Independent | 21 | 20 | 25
  Baseline Independent(n=21,20,25) - 24 mo Dependent | 0 | 0 | 0

18. Secondary Outcome: Change From Baseline in the Number of Infections Requiring Treatment With IV Antibiotics Per Treatment Cycle (28 Days) for the Initial Study Period
Description: Baseline uses the average number of infections requiring IV antibiotic treatment from the 28 days prior to and including the day of first dose to an initial treatment arm. Initial study period values total the number of infections requiring IV antibiotic treatment divided by the number of treatment cycles (each cycle is approximately one month).
Time Frame: 6 months
Population: Intent to treat population
Measure: Median (Full Range); unit: infections per cycle
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5
Number analyzed (Participants) | 50 | 50 | 48
infections per cycle | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 1.00] | 0.00 [-0.89 to 7.00]

19. Secondary Outcome: Change From Baseline in the Number of Infections Requiring Treatment With IV Antibiotics Per Treatment Cycle (28 Days) for the Maintenance Study Period
Description: Baseline uses the average number of infections requiring IV antibiotic treatment from the 28 days prior to and including the day of first dose to an initial treatment arm. Maintenance study period values total the number of infections requiring IV antibiotic treatment divided by the number of treatment cycles (each cycle is approximately one month).
Time Frame: 24 months
Population: Intent to treat population
Measure: Median (Full Range); unit: infections per cycle
Arm/Group | Maintenance Aza 5 Days q 4 Weeks | Maintenance Aza 5 Days q 6 Weeks | Initial Period Treatment Continued Into Maintenance
Number analyzed (Participants) | 22 | 21 | 27
infections per cycle | 0.00 [-1.00 to 0.00] | 0.00 [0.00 to 0.20] | 0.00 [0.00 to 0.67]

ADVERSE EVENTS:
Time Frame: The 3 groups in the Initial Period cover Day 1-6 months, and up to 24 months for participants that continued that treatment. The 2 Maintenance Period groups cover months 7-24 for subjects who were randomized to 1 of the 2 Maintenance treatment arms.
Description: Safety population includes participants who received study treatment. Treatment emergent AEs include events within 42 days of the date of last dose.
Arm/Group | Aza-5 | Aza-5-2-2 | Aza-5-2-5 | Maintenance Aza 5 Days q 4 Weeks | Maintenance Aza 5 Days q 6 Weeks
Serious Adverse Events (participants affected / at risk) | 18/50 | 27/50 | 22/48 | 7/22 | 13/21
Other Adverse Events (participants affected / at risk) | 49/50 | 50/50 | 46/48 | 18/22 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aza-5 (N=50) | Aza-5-2-2 (N=50) | Aza-5-2-5 (N=48) | Maintenance Aza 5 Days q 4 Weeks (N=22) | Maintenance Aza 5 Days q 6 Weeks (N=21)
Anaemia (Blood and lymphatic system disorders) | 2 | 5 | 1 | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 2 | 3 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 2 | 0 | 1
Cardiac valve vegetation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Candida sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fungal oesophagitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Incision site cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 2 | 2 | 1 | 1
Lung infection pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 5 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 4 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 0 | 2 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1 | 2 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Vaginal polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aza-5 (N=50) | Aza-5-2-2 (N=50) | Aza-5-2-5 (N=48) | Maintenance Aza 5 Days q 4 Weeks (N=22) | Maintenance Aza 5 Days q 6 Weeks (N=21)
Anaemia (Blood and lymphatic system disorders) | 11 | 17 | 12 | 3 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 8 | 10 | 9 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 5 | 3 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 15 | 22 | 17 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 14 | 12 | 2 | 5
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 7 | 6 | 0 | 0
Constipation (Gastrointestinal disorders) | 28 | 25 | 21 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 13 | 15 | 14 | 3 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 6 | 3 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 31 | 31 | 23 | 2 | 6
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 4 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 18 | 12 | 13 | 1 | 2
Asthenia (General disorders) | 10 | 8 | 8 | 1 | 4
Chest pain (General disorders) | 1 | 5 | 1 | 1 | 2
Chills (General disorders) | 2 | 3 | 2 | 2 | 2
Fatigue (General disorders) | 25 | 30 | 29 | 5 | 3
Gait disturbance (General disorders) | 0 | 3 | 1 | 0 | 0
Injection site bruising (General disorders) | 11 | 9 | 3 | 1 | 2
Injection site desquamation (General disorders) | 7 | 2 | 3 | 0 | 0
Injection site erythema (General disorders) | 28 | 28 | 26 | 1 | 3
Injection site haemorrhage (General disorders) | 0 | 1 | 4 | 0 | 0
Injection site inflammation (General disorders) | 3 | 1 | 4 | 0 | 0
Injection site nodule (General disorders) | 2 | 1 | 3 | 0 | 0
Injection site pain (General disorders) | 15 | 18 | 18 | 1 | 3
Injection site pruritus (General disorders) | 12 | 6 | 4 | 2 | 1
Injection site rash (General disorders) | 5 | 6 | 4 | 0 | 0
Injection site urticaria (General disorders) | 3 | 1 | 0 | 0 | 0
Injection site warmth (General disorders) | 4 | 2 | 2 | 0 | 0
Oedema peripheral (General disorders) | 4 | 14 | 16 | 3 | 3
Pain (General disorders) | 4 | 1 | 2 | 0 | 0
Pyrexia (General disorders) | 5 | 12 | 10 | 3 | 5
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 3 | 1 | 3 | 0
Oral candidiasis (Infections and infestations) | 0 | 3 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 3 | 3 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 9 | 4 | 6 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 7 | 7 | 7 | 1 | 3
Excoriation (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 3 | 2 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 3 | 0 | 0
Blood urea increased (Investigations) | 1 | 3 | 2 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 4 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 5 | 13 | 6 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2 | 5 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 8 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 5 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 8 | 4 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 4 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 11 | 12 | 11 | 3 | 1
Headache (Nervous system disorders) | 13 | 4 | 7 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 3 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 3 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 3 | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 3 | 2 | 0
Anxiety (Psychiatric disorders) | 3 | 5 | 4 | 0 | 0
Depression (Psychiatric disorders) | 3 | 8 | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 8 | 9 | 5 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 3 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 3 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 4 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 5 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 11 | 9 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 6 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 5 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 3 | 5 | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 8 | 6 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 7 | 2 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 8 | 4 | 0 | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 4 | 6 | 2 | 0 | 3
Pallor (Vascular disorders) | 3 | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present study data provided that the investigator shall (i)furnish the sponsor a copy of any proposed publication or presentation generally thirty (30) days in advance of the submission, (ii) delete any confidential information of the sponsor, and (iii) delay submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner.